CLINICAL TRIAL: NCT01940497
Title: National Phase IIIb Prospective Two-Cohort Non-Randomized, Multi-centre, Open Label Study to Assess the Safety of Subcutaneous Trastuzumab and Molecular Biomarkers in Patients With Early and Locally Advanced HER2-Positive Breast Cancer
Brief Title: A Study of the Safety of Subcutaneously Administered Trastuzumab (Herceptin) in Participants With Early and Locally Advanced Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Acronym: SCHEARLY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ML28879; 2013-001161-16 (EudraCT Number)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trastuzumab (Vial) (Experimental): Participants will receive trastuzumab 600 mg SC using a vial q3w (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
  Interventions: Drug: Doxorubicin; Drug: Docetaxel; Drug: Paclitaxel; Drug: Trastuzumab
- Trastuzumab (SID) (Experimental): Participants will receive trastuzumab 600 mg SC using SID q3w (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
  Interventions: Drug: Doxorubicin; Drug: Docetaxel; Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Doxorubicin — Participants will receive doxorubicin in doses according to the locally-approved regimen q3w (1 cycle), for 4 cycles prior to initiation of trastuzumab treatment.
Drug: Docetaxel — Participants will receive docetaxel in doses according to the locally-approved regimen q3w for 12 weeks, in combination with trastuzumab.
Drug: Paclitaxel — Participants will receive paclitaxel in doses according to the locally-approved regimen weekly for 12 weeks, in combination with trastuzumab.
Drug: Trastuzumab — Participants will receive trastuzumab 600 mg SC (vial or SID) q3w for 18 cycles.
  Other Names: Herceptin

SUMMARY:
This non-randomized, multicenter, open-label study will assess the safety and efficacy of subcutaneously administered trastuzumab in participants with early and locally advanced HER2-positive breast cancer in two sequential cohorts. First 120 participants will be treated with subcutaneous (SC) trastuzumab 600 milligrams (mg) vial (Cohort A) and the subsequent 120 participants will be treated with SC trastuzumab prefilled single use injection device (SID) (Cohort B). Participants from each cohort will receive neoadjuvant or adjuvant chemotherapy consisting of doxorubicin every 3 weeks (q3w) (1 cycle) for 4 cycles followed by paclitaxel weekly or docetaxel every 3 weeks (q3w) in combination with SC trastuzumab (600 mg) q3w for 4 cycles and a further 14 cycles of SC trastuzumab (600 mg) q3w alone. All participants will be followed up for 24 months after the last participant has received the last dose of study treatment, or earlier in case of withdrawal from the study, loss to follow-up or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast. Stage of disease: T1-4 (T describes size of tumour from 1 to 4), N0-3 (N describes nearby lymph nodes), M0 (M describes distant metastasis)
* HER2-positive disease immunohistochemistry (IHC) 3+ or in situ hybridization (ISH) positive
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Left ventricular ejection fraction (LVEF) of greater than or equal to (>=) 55 percent (%) measured by echocardiography (ECHO) or multiple gated acquisition (MUGA) scan prior to first dose of trastuzumab SC
* Intact skin at site of SC injection on the thigh

Exclusion Criteria:

* History of other malignancy, except for participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma and participants with other curatively treated malignancies, other than breast cancer, who have been disease-free for at least 5 years
* Severe dyspnea at rest or requiring supplementary oxygen therapy
* Concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab, specifically: history of documented congestive heart failure (CHF), high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), diagnosed poorly controlled hypertension
* Known infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Pregnant or lactating women
* Concurrent enrolment in another clinical trial using an investigational anti-cancer treatment, including hormonal therapy, bisphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin including hyaluronidase, or the adhesive of the SC device (for Cohort B), or a history of severe allergic or immunological reactions, for example, difficulty to control asthma
* Inadequate bone marrow, hepatic or renal function
* Hormonal treatment concomitant with chemotherapy (allowed in adjuvant phase with adjuvant trastuzumab SC)
* Pre-existing motor or sensory neuropathy of Grade greater than (>) 1
* Synchronous bilateral invasive breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Italy (54):
  - Asl 4 - Osp. San Salvatore; Oncologia Medica, L’Aquila, Abruzzo
  - Ospedale San Carlo; Day Hospital Oncologia Medica, Potenza, Basilicate
  - Campus Universitario S.Venuta; Centro Oncologico T.Campanella, Catanzaro, Calabria
  - Az. Osp. ; Divisione Oncologia Medica, Reggio Calabria, Calabria
  - Azienda Ospedaliera S.G. Moscati; Division of Medical Oncology, Avellino, Campania
  - Presidio Ospedaliero S. Giovanni Di Dio; U.O. Di Oncologia, Frattamaggiore, Campania
  - Seconda Università di Napoli;Day Hospital Clinica Oncologia Medica, Napoli, Campania
  - Ospedale Bellaria; U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Ospedale Ramazzini ; Day Hospital Oncologico, Carpi, Emilia-Romagna
  - Ospedale Civile; Day Hospital Oncologico, Guastalla, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Policlinico A. Gemelli-Complesso Integrato Columbus-Radioterapia, Rome, Lazio
  - Uni Cattolica Policlinico Gemelli; Oncologia Medica Ist. Medicina Interna, Rome, Lazio
  - Ospedale S.G.Calibita Fatebenefratelli; Unità Operativa Oncologia, Rome, Lazio
  - Villa San Pietro Fatebenefatelli; Divisione Oncologia, Rome, Lazio
  - Az. Osp. Uni Ria San Martino; Cliniche Uni Rie Convenzionate U.O. Oncologia Medical, Genoa, Liguria
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Ospedale Civile S. Andrea; Day Hospital Oncologia, La Spezia, Liguria
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Casa Di Cura Poliambulanza; Unita Operativa Di Oncologia Medica, Brescia, Lombardy
  - Ospedale Valduce;U.O.S. Oncologia Ed Ematologia, Como, Lombardy
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - Az. Osp. Carlo Poma; Divisione Di Oncologia Medica, Mantova, Lombardy
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Salvatore Maugeri; Divisione Di Oncologia Medica, Pavia, Lombardy
  - Az. Osp. Di Busto P.O. Di Saronno; U.O. Di Oncologia Medica, Saronno, Lombardy
  - ASST DI BERGAMO OVEST; Unità Operativa di Oncologia Medica, Treviglio, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi; Oncologia Medica, Varese, Lombardy
  - Azienda Sanitaria Locale Di Asti-P.O. Cardinal Massaia;Oncologia, Asti, Piedmont
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Azienda Sanitaria Ospedaliera s. Croce e Carle; Oncologia Medica, Cuneo, Piedmont
  - Ospedale Degli Infermi Di Biella; Reparto Oncologia Medica, Ponderano (BI), Piedmont
  - Ospedale Mauriziano Umberto I; Divisione Onco-Ematologia, Turin, Piedmont
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - A.O.U. Ospedali Riuniti Umberto I-G.M.Lancisi-G.Salesi Ancona;S.O.D. MED.Interna-Clinica Oncologica, Ancona, The Marches
  - Ospedale Di Macerata; Oncologia, Macerata, The Marches
  - Ospedale San Salvatore Muraglia;Divisone Oncologia, Pesaro, The Marches
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Ospedale della Misericordia; Hospice Terapia del Dolore, Grosseto, Tuscany
  - Ospedale Nuovo Della Versilia; Divisione Di Oncologia Medica, Lido di Camaiore, Tuscany
  - Ospedale Civile; Unita Operativa Di Oncologia Medica, Livorno, Tuscany
  - Azienda Usl 7; Dept. Oncologico, Poggibonsi, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Sant'Andrea Delle Fratte (PG), Umbria
  - Presidio Ospedaliero - Usl 13; Servizio Di Oncologia, Castelfranco Veneto, Veneto
  - AZ. Usll12 Veneziana-Ospedale Dell'angelo;Oncologia Medica, Mestre, Veneto
  - Ospedale Calvi di Noale; U.O. Complessa di Oncologia ed Ematologia Oncologica, Mirano, Veneto
  - Ospedale Sacro Cuore Don Calabria; U.O. Di Oncologia, Negrar, Veneto
  - Ospedale Cà Foncello - Divisione di Oncologia Medica, Treviso, Veneto
  - Ospedale Di Vicenza; Nefrologia, Oncologia Medica, Vicenza, Veneto

REFERENCES:
- [Derived] Zambetti M, Montemurro F, Morandi P, Zamagni C, Brandes AA, Bisagni G, Cagossi K, Bengala C, Gori S, Iannacone C, Stell A, Gianni L. Safety profile of subcutaneous trastuzumab for the treatment of patients with HER2-positive early or locally advanced breast cancer: primary analysis of the SCHEARLY study. Eur J Cancer. 2018 Dec;105:61-70. doi: 10.1016/j.ejca.2018.09.034. Epub 2018 Nov 3. PMID 30396014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 263 screened participants, 240 participants were enrolled in the study.
Groups:
- Trastuzumab (Vial): Participants received trastuzumab 600 milligrams (mg) subcutaneously using a vial every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (SID): Participants received trastuzumab 600 mg subcutaneously using single-use injection device (SID) every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
Period: Overall Study
Arm/Group | Trastuzumab (Vial) | Trastuzumab (SID)
Started | 121 | 119
Treated | 115 | 113
Treated: Adjuvant | 95 | 92
Treated: Neoadjuvant | 20 | 21
Completed (Completed Treatment Period) | 100 | 101
Not Completed | 21 | 18
Not completed — Adverse Event/Intercurrent Illness | 11 | 8
Not completed — Recurrence of Disease Postsurgery | 1 | 3
Not completed — Violation of Entry Criteria | 1 | 1
Not completed — Refused Treatment | 1 | 3
Not completed — Withdrew Consent | 6 | 2
Not completed — Administrative/Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab (Vial) | Trastuzumab (SID) | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.51) | 53.2 (10.37) | 54.2 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 119 | 239
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were the AEs occurring from starting on the day of or after first administration of trastuzumab and within 28 days after last dose of trastuzumab. Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: Day 1 up to 28 days after last dose of trastuzumab (up to approximately 1 year)
Population: Safety population
Measure: Number; unit: Percentage of Participants
Groups:
- Trastuzumab (Vial): Adjuvant: Participants received trastuzumab 600 mg subcutaneously using a vial every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (Vial): Neoadjuvant: Participants received trastuzumab 600 mg subcutaneously using a vial every 3 weeks (1 cycle) for 1 year (4 cycles in combination with neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (SID): Adjuvant: Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (SID): Neoadjuvant: Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 95 | 20 | 92 | 21
Percentage of Participants | 98.9 | 100.0 | 89.1 | 95.2

2. Secondary Outcome: Actual Dose of Trastuzumab Administered
Description: Actual dose (mg) administered = (sum over all cycles of actual dose received [mg] divided by number of cycles). Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: Day 1 up last dose of trastuzumab (up to approximately 1 year)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 95 | 20 | 92 | 21
mg | 599.7 (3.08) | 600.00 (0.000) | 593.3 (16.55) | 595.9 (10.4)

3. Secondary Outcome: Duration of Treatment With Trastuzumab
Description: Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: Day 1 up last dose of trastuzumab (up to approximately 1 year)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 95 | 20 | 92 | 21
days | 346 (72.13) | 352.2 (55.82) | 340.1 (85.47) | 351.9 (90.02)

4. Secondary Outcome: Percentage of Participants Who Received Concomitant Medications
Time Frame: Screening (Day -28 to -1) up to 2.5 years
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Groups:
- Trastuzumab (Vial): Participants received trastuzumab 600 mg subcutaneously using a vial every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (SID): Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
Arm/Group | Trastuzumab (Vial) | Trastuzumab (SID)
Number analyzed (Participants) | 115 | 113
Percentage of Participants | 100 | 100

5. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR) (Neoadjuvant Groups Only) Using Mammography
Description: In the neoadjuvant setting, the activity of two sequential drug regimens, doxorubicin-containing chemotherapy followed by paclitaxel or docetaxel chemotherapy in combination with trastuzumab, was assessed as the percentage of participants with pCR in breast and nodes using mammography. pCR was defined as the absence of histological evidence of invasive breast cancer cells in the tissue specimen removed from the breast after preoperative treatment. Data for this outcome measure were analyzed and reported only for neoadjuvant groups within each treatment arm.
Time Frame: Day 1 up to 24 weeks
Population: Modified intent-to-treat (m-ITT) population included all enrolled participants satisfying criteria for eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 22 | 19
Percentage of Participants | 40.9 [31.0 to 51.0] | 15.8 [8.00 to 24.0]

6. Secondary Outcome: Percentage of Participants With Event (Local, Regional or Distant Recurrence, Contralateral Breast Cancer or Death) Using Mammography
Description: A participant was considered as disease free if the participant was free from local, regional or distant recurrence, contralateral breast cancer or death due to any cause (whichever occurred first). Percentage of participants with event at the cut off date were reported. Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: Day 1 up to local, regional or distant recurrence, contralateral breast cancer or death due to any cause (whichever occurred first [up to approximately 4.5 years])
Population: m-ITT population. Here, 'Number of Participants Analyzed' = participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 92 | 18 | 91 | 18
Percentage of Participants | 18.5 | 33.3 | 6.6 | 11.1

7. Secondary Outcome: Disease-Free Survival (DFS) Using Mammography
Description: DFS was defined as the time from the first treatment to local, regional or distant recurrence, contralateral breast cancer or death due to any cause (whichever occurred first). Kaplan-Meier estimates were used for analysis. Participants who were disease-free were censored at the data cut off date. Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: as for outcome 6
Population: m-ITT population. Here, 'Number of Participants Analyzed' = participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 92 | 18 | 91 | 18
Months | NA [NA to NA] — Median and corresponding 95% confidence interval (CI) could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date.

8. Secondary Outcome: Percentage of Participants Who Died
Description: as for outcome 3
Time Frame: Day 1 up to death due to any cause (up to approximately 4.5 years)
Population: m-ITT population
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 96 | 22 | 93 | 19
Percentage of Participants | 5.2 | 4.5 | 0.0 | 5.26

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the first treatment to death from any cause. Kaplan-Meier estimates were used for analysis. Participants who did not die were censored on the date they were last known to be alive. Data for this outcome measure were analyzed and reported by adjuvant versus neoadjuvant chemotherapy groups within each treatment arm.
Time Frame: Day 1 up to death due to any cause (up to approximately 4.5 years)
Population: m-ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID): Adjuvant | Trastuzumab (SID): Neoadjuvant
Number analyzed (Participants) | 96 | 22 | 93 | 19
Months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated because majority of participants were censored at data cut off date.

10. Secondary Outcome: Percentage of Participants by Response to Patient Satisfaction Questionnaire (PSQ)
Description: Participants were asked the following 5 questions: (1) "Following the first injection given by the physician/nurse and training on how to use the SID, I felt comfortable injecting the study drug by myself"; (2) "The SID was convenient and easy to use"; (3) "I am confident giving myself an injection in the thigh with the SID"; (4) "Taking all things into account, I find self-administration using the SID satisfactory"; (5) "If given the opportunity, I would choose to continue self-injecting the study drug using the SID at home". Response to each question was recorded as either of the following options: "Unknown", "Strongly Disagree", "Disagree", "Unsure", "Agree", "Strongly Agree". Percentage of participants who provided responses to above questions was reported. Data for this outcome measure were analyzed and reported only for Trastuzumab (SID) arm.
Time Frame: After at least 14 cycles (1 cycle = 21 days; maximum up to 1 year)
Population: PSQ population included all enrolled participants from trastuzumab (SID) group who were able to use SID and had completed a minimum of 14 administrations of trastuzumab subcutaneously using SID (at least 10 of which were self-administered). Here, 'Number of Participants Analyzed' = participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab (SID)
Number analyzed (Participants) | 15
Percentage of Participants
  Comfortable: Unknown | 0.0
  Comfortable: Strongly Disagree | 0.0
  Comfortable: Disagree | 0.0
  Comfortable: Unsure | 6.7
  Comfortable: Agree | 40
  Comfortable: Strongly Agree | 53.3
  Convenient: Unknown | 0.0
  Convenient: Strongly Disagree | 0.0
  Convenient: Disagree | 0.0
  Convenient: Unsure | 6.7
  Convenient: Agree | 33.3
  Convenient: Strongly Agree | 60
  Confident: Unknown | 0.0
  Confident: Strongly Disagree | 0.0
  Confident: Disagree | 0.0
  Confident: Unsure | 6.7
  Confident: Agree | 40.0
  Confident: Strongly Agree | 53.3
  Satisfactory: Unknown | 0.0
  Satisfactory: Strongly Disagree | 0.0
  Satisfactory: Disagree | 0.0
  Satisfactory: Unsure | 6.7
  Satisfactory: Agree | 33.3
  Satisfactory: Strongly Agree | 60
  Would continue: Unknown | 0.0
  Would continue: Strongly Disagree | 0.0
  Would continue: Disagree | 13.3
  Would continue: Unsure | 6.7
  Would continue: Agree | 20
  Would continue: Strongly Agree | 60

11. Secondary Outcome: Percentage of Health Care Professionals (HCPs) by Response to Health Care Professional Questionnaire (HCPQ)
Description: Percentage of HCPs providing responses to various questions related to overall ease of study drug administration was reported in different categories, where categories indicate all possible responses to such questions.
Time Frame: After at least 4 participants completed 5 cycles of adjuvant treatment (1 cycle = 21 days; maximum up to 1 year)
Population: HCPQ population included all investigators and study nurses who completed the questionnaire at each site when at least 4 participants from their site had received at least 5 cycles of adjuvant study treatment (52 and 50, respectively for Vial and SID groups).
Measure: Number; unit: Percentage of HCPs
Groups:
- HCPs: Trastuzumab (Vial): Participants received trastuzumab 600 mg subcutaneously using a vial every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone). Trastuzumab using vial had to be administered by an HCP.
- HCPs: Trastuzumab (SID): Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant or neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone). Trastuzumab using SID had to be administered by an HCP or by the participant after appropriate training and under HCP supervision.
Arm/Group | HCPs: Trastuzumab (Vial) | HCPs: Trastuzumab (SID)
Number analyzed (Participants) | 52 | 50
Percentage of HCPs
  Specialization: Oncologist | 17.3 | 16.0
  Specialization: Specialist nurse | 69.2 | 76.0
  Specialization: Other | 11.5 | 8.0
  Specialization: Missing | 1.9 | 0.0
  Personally administered/supervised: Always | 40.4 | 48.0
  Personally administered/supervised: Sometimes | 51.9 | 48.0
  Personally administered/supervised: Never | 7.7 | 4.0
  If 'Never', who administered: Specialist nurse | 7.7 | 4.0
  Syringe prepared at: Pharmacy | 55.8 | NA — Data were not evaluable as this question applied only to vial group.
  Syringe prepared at: Oncology ward | 40.4 | NA — Data were not evaluable as this question applied only to vial group.
  Syringe prepared at: Missing | 3.8 | NA — Data were not evaluable as this question applied only to vial group.
  Time to fill syringe: less than (<) 5 minutes | 67.3 | NA — Data were not evaluable as this question applied only to vial group.
  Time to fill syringe: 6-10 minutes | 13.5 | NA — Data were not evaluable as this question applied only to vial group.
  Time to fill syringe: 11-15 minutes | 5.8 | NA — Data were not evaluable as this question applied only to vial group.
  Time to fill syringe: Unknown | 13.5 | NA — Data were not evaluable as this question applied only to vial group.
  Total time for vial administration: <3 minutes | 1.9 | NA — Data were not evaluable as this question applied only to vial group.
  Total time for vial administration: <5 minutes | 59.6 | NA — Data were not evaluable as this question applied only to vial group.
  Total time for vial administration: 6-15 minutes | 38.5 | NA — Data were not evaluable as this question applied only to vial group.
  Time to prepare SID: <5 minutes | NA — Data were not evaluable as this question applied only to SID group. | 72.0
  Time to prepare SID: 6-10 minutes | NA — Data were not evaluable as this question applied only to SID group. | 14.0
  Time to prepare SID: 11-15 minutes | NA — Data were not evaluable as this question applied only to SID group. | 4.0
  Time to prepare SID: 16-20 minutes | NA — Data were not evaluable as this question applied only to SID group. | 2.0
  Time to prepare SID: >20 minutes | NA — Data were not evaluable as this question applied only to SID group. | 8.0
  Total time for SID administration: <3 minutes | NA — Data were not evaluable as this question applied only to SID group. | 26.0
  Total time for SID administration: <5 minutes | NA — Data were not evaluable as this question applied only to SID group. | 30.0
  Total time for SID administration: 6-15 minutes | NA — Data were not evaluable as this question applied only to SID group. | 44.0
  Injection site: Irritation: A lot | 1.9 | 4.0
  Injection site: Irritation: A few | 46.2 | 36.0
  Injection site: Irritation: None | 51.9 | 60.0
  Injection site: Bruising: A few | 7.7 | 10.0
  Injection site: Bruising: None | 92.3 | 90.0
  Injection site: Infection: None | 100.0 | 100.0
  Fever,shivering,flu-like,rash,swelling:A few | 15.4 | 14.0
  Fever,shivering,flu-like,rash,swelling:None | 84.6 | 86.0
  Time at hospital for administration: <2 hours | 44.2 | 44.0
  Time at hospital for administration: >2, <3 hours | 23.1 | 34.0
  Time at hospital for administration: >3, <4 hours | 23.1 | 12.0
  Time at hospital for administration: >4 hours | 7.7 | 10.0
  Time at hospital for administration: Missing | 1.9 | 0.0
  Anxiety to participants: None | 82.7 | 90.0
  Anxiety to participants: A fair amount | 17.3 | 10.0
  Ease of vial administration: None | 5.8 | NA — Data were not evaluable as this question applied only to vial group.
  Ease of vial administration: A fair amount | 38.5 | NA — Data were not evaluable as this question applied only to vial group.
  Ease of vial administration: A lot | 55.8 | NA — Data were not evaluable as this question applied only to vial group.
  Subcutaneous route may simplify management: Yes | 94.2 | 100.0
  Subcutaneous route may simplify management: No | 5.8 | 0.0
  Would recommend SID to intravenous route: Yes | 96.2 | 96.0
  Would recommend SID to intravenous route: No | 3.8 | 4.0
  Would recommend subcutaneous route to medics: Yes | 100.0 | 90.0
  Would recommend subcutaneous route to medics: No | 0.0 | 8.0
  Would recommend subcutaneous to medics:Missing | 0.0 | 2.0
  Convenience of using SID by participants: Yes | 94.2 | 96.0
  Convenience of using SID by participants: No | 0.0 | 4.0
  Convenience of using SID by participants: Missing | 5.8 | 0.0

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of trastuzumab
Description: Safety population TEAEs
Groups:
- Trastuzumab (SID) Adjuvant: Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with adjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
- Trastuzumab (SID) Neoadjuvant: Participants received trastuzumab 600 mg subcutaneously using SID every 3 weeks (1 cycle) for 1 year (4 cycles in combination with neoadjuvant chemotherapy [consisting of doxorubicin, paclitaxel or docetaxel] and 14 cycles administered alone).
Arm/Group | Trastuzumab (Vial): Adjuvant | Trastuzumab (Vial): Neoadjuvant | Trastuzumab (SID) Adjuvant | Trastuzumab (SID) Neoadjuvant
All-Cause Mortality (participants affected / at risk) | 5/95 | 1/20 | 0/92 | 1/21
Serious Adverse Events (participants affected / at risk) | 5/95 | 3/20 | 7/92 | 2/21
Other Adverse Events (participants affected / at risk) | 92/95 | 20/20 | 79/92 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (Vial): Adjuvant (N=95) | Trastuzumab (Vial): Neoadjuvant (N=20) | Trastuzumab (SID) Adjuvant (N=92) | Trastuzumab (SID) Neoadjuvant (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pryexia (General disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (Vial): Adjuvant (N=95) | Trastuzumab (Vial): Neoadjuvant (N=20) | Trastuzumab (SID) Adjuvant (N=92) | Trastuzumab (SID) Neoadjuvant (N=21)
Neutropenia (Blood and lymphatic system disorders) | 20 | 4 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 15 | 2 | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 10 | 3 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 25 | 3 | 15 | 6
Nausea (Gastrointestinal disorders) | 8 | 2 | 13 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 3 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1 | 5 | 0
Constipation (Gastrointestinal disorders) | 8 | 0 | 7 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 0 | 4 | 0
Asthenia (General disorders) | 32 | 3 | 20 | 7
Pyrexia (General disorders) | 18 | 4 | 13 | 4
Fatigue (General disorders) | 12 | 0 | 12 | 1
Oedema peripheral (General disorders) | 10 | 0 | 11 | 1
Mucosal inflammation (General disorders) | 9 | 0 | 7 | 1
Chest pain (General disorders) | 6 | 1 | 0 | 1
Pain (General disorders) | 7 | 0 | 3 | 1
Influenza like illness (General disorders) | 5 | 1 | 2 | 1
Oedema (General disorders) | 6 | 0 | 2 | 0
Cystitis (Infections and infestations) | 7 | 0 | 8 | 1
Influenza (Infections and infestations) | 3 | 1 | 9 | 3
Ejection fraction decreased (Investigations) | 13 | 2 | 3 | 3
Neutrophil count decreased (Investigations) | 3 | 0 | 6 | 2
White blood cell count decreased (Investigations) | 2 | 0 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 4 | 28 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 0 | 8 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 0 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 8 | 1
Paraesthesia (Nervous system disorders) | 49 | 3 | 25 | 3
Headache (Nervous system disorders) | 6 | 2 | 4 | 1
Dysgeusia (Nervous system disorders) | 6 | 0 | 6 | 1
Neurotoxicity (Nervous system disorders) | 3 | 3 | 5 | 1
Amenorrhoea (Reproductive system and breast disorders) | 4 | 0 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 15 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | 8 | 2
Erythema (Skin and subcutaneous tissue disorders) | 23 | 2 | 14 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 11 | 2 | 9 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 7 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 7 | 0
Hot flush (Vascular disorders) | 7 | 5 | 7 | 2
Hypertension (Vascular disorders) | 7 | 5 | 8 | 1
Lymphoedema (Vascular disorders) | 5 | 1 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 6 | 0 | 1 | 2
Eye disorder (Eye disorders) | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 5 | 0
Injection site erythema (General disorders) | 1 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 3 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 3 | 2 | 2 | 2
Pharyngitis (Infections and infestations) | 3 | 2 | 4 | 1
Mastitis (Infections and infestations) | 2 | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0
Hepatitis C virus test positive (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 2 | 0 | 3 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 5 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 5 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 5 | 0 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 3 | 2 | 5 | 0
Dysuria (Renal and urinary disorders) | 3 | 1 | 4 | 0
Panic attack (Psychiatric disorders) | 1 | 1 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT01940497/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT01940497/SAP_001.pdf